CLINICAL TRIAL: NCT06974812
Title: A Phase 1/2 Study of IBI3014 in Participants With Unresectable Locally Advanced or Metastatic Solid Tumors
Brief Title: IBI3014 in Participants With Unresectable Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI3014A101
Record Dates: First submitted 2025-04-23; First posted 2025-05-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Unresectable Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI3014 (Experimental): IBI3014 will be dosed until disease progression, toxicity intolerance, starting of new systemic anti-cancer treatment, withdrawal of consent, occurrence of other reasons for discontinuing study therapy, or treatment duration reaching the maximum of 24 months, whichever occurs first.
  Interventions: Drug: IBI3014

INTERVENTIONS:
Drug: IBI3014 — 12 mg/kg D1 IV Q3W
Drug: IBI3014 — 6 mg/kg D1 IV Q3W
Drug: IBI3014 — 1 mg/kg D1 IV Q3W
Drug: IBI3014 — 15 mg/kg D1 IV Q3W
Drug: IBI3014 — 9 mg/kg D1 IV Q3W
Drug: IBI3014 — 3 mg/kg D1 IV Q3W
Drug: IBI3014 — 20 mg/kg D1 IV Q3W
Drug: IBI3014 — 18 mg/kg D1 IV Q3W

SUMMARY:
This is a phase 1/2 multicenter, multi-regional, open-label, first-in-human study of IBI3014 in participants with unresectable locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria

* 1.Participants with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
* 2.Male or female participants ≥ 18 years old;
* 3.Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;
* 4.Anticipated life expectancy of ≥ 12 weeks;
* 5.Participants, both male and female, who are either not of childbearing potential or who agree to use at least one highly effective method of contraception during the study (begin from screening or within 2 weeks prior to the first dose, whichever comes first, and continue until 6 months after the last dose of study drug).
* 6.Adequate bone marrow and organ function:
* 7.Has at least 1 measurable lesion per RECIST v1.1(at least 1 evaluable lesion for dose participants in dose escalation part);
* 8.Not a candidate for curable surgical resection or radical chemoradiation;

Exclusion Criteria

* 1.Drugs and other treatments to be excluded;
* 2.Has adverse reactions resulting from previous anti-tumor therapies, which have not resolved to Grade 0 or 1 toxicity according to NCI-CTCAE v5.0 (except for alopecia, fatigue, pigmentation and other conditions with no safety risk according to Investigators' opinion) prior to first administration of the study drug;
* 3.Prior use of Camptothecin-Derived agents (e.g., irinotecan, topotecan) or immune checkpoint inhibitor and documented adverse reaction which is severe and influence the safety assessment of participants.
* 4.Allergic or hypersensitive to other monoclonal antibodies and/or Camptothecin Derivative based therapy, or any ingredients of IBI3014;
* 5.Known symptomatic central nervous system (CNS) metastases. The following conditions could be considered enrollment: Participants with asymptomatic CNS metastases (which means no neural system syndromes, no need of corticosteroids treatment and diameter of metastases ≤ 1.5cm) or confirmed stable status according to Investigators' opinion after treatment, No midbrain, pons, cerebellum, meninges, medulla oblongata or spinal cord metastasis; and stable status for at least 4 weeks without new or enlarged metastases definitively confirmed by clinical evidence, and withdrawal of corticosteroids or anticonvulsant for at least 2 weeks prior to the first administration of study drug;
* 6.History of pneumonitis requiring corticosteroids therapy, or history of clinically significant lung diseases (e.g. Interstitial lung disease, non-infectious pneumonia, or uncontrolled lung disease such as pulmonary fibrosis, severe radiation pneumonitis and acute lung injury) or who are suspected to have these diseases by imaging at screening period;
* 7.Participants with a clinically significant (CS) cardiovascular disease or condition;
* 8.Participants with a significant gastrointestinal disease or condition,
* 9.Participants with biliary obstruction. Unless the blockage is treated locally, such as endoscopic stenting or percutaneous liver puncture and drainage, the total bilirubin is reduced below 1.5 times ULN;
* 10.Ascites, pleural effusion, or pericardial effusion with symptoms and requiring intervention;
* 11.Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh grade B or more severe cirrhosis;
* 12.Significant malnutrition, such as the need for intravenous fluids; Malnutrition corrected for more than 4 weeks prior to the first administration of study drug is allowed;
* 13.Tumor invasion of surrounding important structures (such as mediastinal vessels, superior vena cava, trachea, esophagus, etc.) or at risk of gastrointestinal/respiratory fistula;
* 14.Uncontrolled or clinically significant infections
* 15.History of immunodeficiency disease, including congenital or acquired immunodeficiency diseases;
* 16.Had a history of organ transplantation, allogeneic bone marrow transplantation or hematopoietic stem cell transplantation;
* 17.Other uncontrolled active disease or acute or chronic diseases or abnormal laboratory test that may: increase risk of study participation or study drug administration, interfere with the interpretation of study results, and, disqualify the participant for study participation in the Investigator's judgment;
* 18.History of other primary malignant tumors;
* 19.Women who are considered pregnant or are lactating;
* 20.Under neurological, psychiatric disorder or social condition that affects compliance with study requirements, significantly increases the risk of adverse events, or affects participants' ability to provide written informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The Safety profile of patients in Phase 1 dose escalation part、Phase 1 dose expansion and Phase 2 dose optimization | 2 years after LPI
  Number ofparticipants with adverse events (AEs)
Dose limiting toxicity (DLT) of IBI3014 in Phase 1 dose escalation | 21 days after LPI
  The occurance of Dose limiting toxicity (DLT) per protocol to establish MTD or RDEs
ORR per RECIST v1.1 in Phase 1 dose expansion and Phase 2 dose optimization | 2 years after LPI
  The investigator assessed ORR per RECIST v1.1
The Safety profile of patients in Phase 1 dose escalation part、Phase 1 dose expansion and Phase 2 dose optimization | 2 years after LPI
  Number ofparticipants with abnormal laboratorytests results
The Safety profile of patients in Phase 1 dose escalation part、Phase 1 dose expansion and Phase 2 dose optimization | 2 years after LPI
  Number ofparticipants with abnormal physical examination findings
The Safety profile of patients in Phase 1 dose escalation part、Phase 1 dose expansion and Phase 2 dose optimization | 2 years after LPI
  Number ofparticipants with abnormal vital signs

SECONDARY OUTCOMES:
Efficacy of IBI3014 | 2 years after LPI
  DOR, DoR, TTR, PFS as evaluated by investigator per RECIST v1.1 criteria and OS
PK profile of IBI3014 | 2 years after LPI
  area under the curve (AUC)
Incidence and characterization of anti-IBI3014 antibodies | 2 years after LPI
  Rate of ADA and Nab
PK profile of IBI3014 | 2 years after LPI
  area under the Cmax
PK profile of IBI3014 | 2 years after LPI
  area under the Tmax
PK profile of IBI3014 | 2 years after LPI
  area under the Clearance
PK profile of IBI3014 | 2 years after LPI
  area under the t1/2 and others

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian cancer hospital, Fuzhou, Fujian
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality